# **Study Protocol**

Official Title: Erectile Dysfunction and the Mind: Evaluating the Influence of

Depression and Illness Beliefs on Treatment Progression

NCT Number: NCT06996925

Document Date: August 6, 2025

Institution: Haseki Training and Research Hospital

Principal Investigator: Nazım Furkan Günay

Email: nfurkangunay@gmail.com

# 1. Background and Rationale

Erectile dysfunction (ED) is a complex and multifactorial condition...

# 2. Objectives

Primary Objective: To assess the association between illness perception and depressive symptoms in ED patients.

Secondary Objectives: To evaluate changes in erectile function and depression over 1 month.

## 3. Study Design

Study Type: Observational

Model: Cohort

Time Perspective: Prospective

Number of Cohorts: 1

Target Follow-Up Duration: 1 month

Enrollment: 120 participants anticipated

Biospecimen Retention: None Retained

## 4. Study Population

**Inclusion Criteria:** 

- Male, aged 18 or older
- Diagnosed with ED
- Consent to participate

#### **Exclusion Criteria:**

- Severe psychiatric disorder
- Hormonal or cancer therapy
- Neurological diseases

### 5. Procedures

Patients will complete IIEF-5, B-IPQ, and PHQ-9 at baseline and at 1-month follow-up.

### 6. Statistical Considerations:

Descriptive statistics will be used to summarize baseline characteristics. Paired t-tests or Wilcoxon signed-rank tests will be used to compare baseline and follow-up scores. A p-value < 0.05 will be considered statistically significant.

### 7. Ethical Considerations

This study was approved by the Ethics Committee of Haseki Training and Research Hospital on March 19, 2025 (Approval No: 23-2025). No amendments were made to the original protocol before submission. The current version has been approved by the ethics committee.

## 8. Data Management

CRFs and SOPs will guide data entry, quality checks, and confidentiality procedures.